CLINICAL TRIAL: NCT02909374
Title: "Stay Balanced" - Prevention of Falls in Older Adults Through Implementation of Evidence Based Balance Training - From Clinical Research to Clinical Practice
Brief Title: "Stay Balanced" - Prevention of Falls in Older Adults - From Clinical Research to Clinical Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Alexandra Halvarsson, medicine doctor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Dnr 2016/415-31
Record Dates: First submitted 2016-04-06; First posted 2016-09-21 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Prevention Harmful Effects
Keywords: Implementation; fall prevention; balance training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance training (Experimental): The program includes exercise with dual- and multi task performance and is progressive as the exercises can be performed at different levels (basic, moderate, and advanced). The 12-week balance training program will be performed two times per week for one hour each. The training will be lead by physiotherapists or trained leaders. After the balance training the participants will get recommendations for continued physical activity and training, i.e. "Physical activity on prescription".
  Interventions: Other: Balance training

INTERVENTIONS:
Other: Balance training — The balance-training program was developed based on well-established principles of exercise and on the knowledge that balance control relies on the interaction of several physiological systems, as well as interaction with environmental factors and the performed task. It includes exercise with dual- and multi task performance. It is progressive as the exercises can be performed at different levels (basic, moderate, and advanced), making it progressively challenging for each individual throughout the whole program. The training is conducted as an individually tailored group program.

SUMMARY:
Fall is one of the most common causes of ill health and morbidity in the older population. In Sweden about 300 000 people/year seek emergency treatment due to falls and out of these 1600 dies. Poor balance control leads to a sedentary life with muscle weakness, fear of falling and an increased risk for falls. Balance training and physical activity have positive effects on fall prevention and balance, but long-term follow-ups are limited. There is also a gap between what has been proven to be efficient in research and what is performed in communities and clinical settings.

Many studies reports on the efficacy of certain treatment, method or training program, which often may have taken years to develop, but few of these results are taken further into clinical practice and it may take years for them to come into daily use. This delay means that there is a gap between what is known and what is consistently done. It if of importance implement methods that have been proven to have beneficial impact on health and physical function in a clinical trial. Furthermore to evaluate which strategies for implementation that are of significance. The aim of this study is to implement evidence based balance training into clinical practice to prevent future falls and fall-related injuries in older adults.

The program has been proven to be efficient, but not yet been implemented in the community and clinical settings. Implementation outcomes will include effectiveness, acceptability, feasibility, fidelity, cost and sustainability. Outcome variables on individual level will be fall-related concerns, balance performance, physical function and activity, health related quality of life and number of falls.

The investigators foresee that this balance training for older adults will prevent future falls and fall related injuries, increase physical activity level, health related quality of life and provide the participants with a strategy to be able to have a physically active and healthy life style.

DETAILED DESCRIPTION:
This project is a cluster-randomized study comparing different implementation strategies. The study will comprise clinical settings in primary health care (PHC) and in senior residential care.

Participating clinics will be recruited strategically with regard to catchment area and population structure, to achieve such a large diverse participation as possible.

Participant to the balance training will be recruited through the participating clinics, from primary care facilities in the vicinity of the clinics involved and by advertisement in local papers in the communities. Participants reporting their interest to partake in the study will be telephone-interview and informed about the project and checked for eligibility. Thereafter, they will be called to baseline testing.

The investigators plan to involve 30 different PHC and thereby 360-480 participants in balance training (two groups with 6-8 participants per semester from each clinic during 2 semesters).

In two previous randomised controlled studies performed by the research group in Stockholm county regarding group balance-training for older adults at risk of falling the investigators received a large number of people reporting interest by announcement, i.e. approximately 500 subjects. However, most of them were excluded because they had not a verified diagnosis of osteoporosis, which was one of the inclusion criteria's in those two studies.

The group based balance-training program is well described in a published ´Rehabilitation in practice´- article and was developed based on well-established principles of exercise and on the knowledge that balance control relies on the interaction of several physiological systems, as well as interaction with environmental factors and the performed task. It includes exercise with dual- and multi task performance, i.e. performance when a person's attention is divided between a motor and a cognitive task, as this is a natural component of daily activities, but may increase the risk of falling especially in older adults. As training adaptions are specific for the system trained, this program follows the principle of specificity in that it is based on exercises targeting various systems for postural control aiming to improve balance performance in specific situations that can occur in daily life, such as regaining postural stability after perturbation or being able to suddenly avoid an obstacle, with retained balance, while simultaneously walking and answering a question. Furthermore, it is progressive as the exercises can be performed at different levels (basic, moderate, and advanced), making it progressively challenging for each individual throughout the whole program. The training is conducted as an individually tailored group program. The 12-week balance training program will be performed two times per week for one hour each. The training will be lead by physiotherapists or trained leaders. After the balance training the participants will get recommendations for continued physical activity and training, i.e. "Physical activity on prescription".

For the implementation a participatory approach will be used, where the different settings will be engaged in an early phase. For evaluation the model by Proctor et al., will be followed. The implementation strategies will include 1) a contract with each setting, 2) meetings with the head of each setting, 3) discussion with physical therapists and leaders in the setting, 4) education of the physical therapists and leaders who will be trainers and 5) coaching of the trainers.

Implementation outcomes will include:

* Acceptability of evidence-based treatments among health providers will be assessed by investigating the attitudes towards the balance program with a questionnaire, focus groups and interviews.
* Feasibility the extent to which a new treatment can be successfully used and carried out in the clinical setting will be assessed by investigating how the balance program fits in in clinical practice with focus groups and interviews.
* Fidelity includes five dimensions, i.e. adherence to the program protocol, quality of delivery, program component differentiation, exposure to the intervention and participant responsiveness to the program will be investigated by observations, check-lists and assessments on individual level (see below).
* Cost will be assessed by a health economic evaluation of the program.
* Sustainability will be assessed using both quantitative and qualitative methods and include measures on compliance/fidelity to the training program.

Assessments on individual level will include fall-related concerns, health related quality of life, balance performance, gait, physical activity, muscle strength for lower extremities and number of falls and compliance to training.

The assessments on individual level will be performed at the PHC by the regular physiotherapist. All participants will be assessed before and after the training period (3 months after inclusion) and at three to six, twelve eight-teen and twenty-four months, i.e. two years after inclusion. During the follow-up period, i.e. three, six, twelve, eight-teen and twenty-four months, the assessments will consists of sms-track system and by postal survey with questionnaire regarding fall-related concerns, heath related quality of life, physical activity and adherence to training regime.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older, independent ambulatory indoors, self-perceived balance problems and/or fear of falling.

Exclusion Criteria:

* Had fall-related fractures during the last six months,
* Severely decreased vision, or other diseases or constrains that might interfere with participation in the training program.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Sustainability of the balance training programme in clinical setting | Sustainability will be assessed during a period of 18 months
  Sustainability will be assessed using both quantitative and qualitative methods and include measures on compliance/fidelity to the training program. A successful implementation will be consider if the clinic has contained/sustained the balance training during 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Halvarsson, med.dr, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Halvarsson A, Roaldsen KS, Nilsen P, Dohrn IM, Stahle A. StayBalanced: implementation of evidence-based fall prevention balance training for older adults-cluster randomized controlled and hybrid type 3 trial. Trials. 2021 Feb 26;22(1):166. doi: 10.1186/s13063-021-05091-1. PMID 33637122